CLINICAL TRIAL: NCT03927456
Title: A Phase III Study to Evaluate the Efficacy and Safety of SHR6390 in Combination With Fulvestrant Versus Placebo Combined With Fulvesrant in Patients With HR Positive and HER2 Negative Recurrent/Metastatic Breast Cancer
Brief Title: A Study of SHR6390 in Combination With Fulvestrant in Patients With HR Positive and HER2 Negative Advanced Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR6390-III-301
Record Dates: First submitted 2019-04-17; First posted 2019-04-25 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2020-06

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR6390 + Fulvestrant (Experimental): Intervention Drug: SHR6390, Fulvestrant
  Interventions: Drug: SHR6390; Drug: Fulvestrant
- Placebo + Fulvestrant (Placebo Comparator): Intervention Drug: Placebo, Fulvestrant
  Interventions: Drug: Placebo; Drug: Fulvestrant

INTERVENTIONS:
Drug: SHR6390 — SHR6390 150 mg, orally once daily on Day 1 to Day 21 of every 28-day cycle followed by 7 days off treatment
  Arms: SHR6390 + Fulvestrant
Drug: Placebo — Placebo 150 mg, orally once daily on Day 1 to Day 21 of every 28-day cycle followed by 7 days off treatment
  Arms: Placebo + Fulvestrant
Drug: Fulvestrant — Fulvestrant 500mg intramuscular injection on day 1 and day 15 for the first cycle and then on day 1 for every cycle until progressive disease

SUMMARY:
This is a phase III clinical trial to evaluate the efficacy and safety of SHR6390 in combination with Fulvestrant versus placebo combined with Fulvesrant in Patients who have HR positive and HER2 negative recurrent/metastatic breast cancer and have received prior endocrine therapy are eligible for study.

ELIGIBILITY:
Inclusion Criteria:

1. Has the pathologically-confirmed diagnosis of locally recurrent or metastatic, hormone-receptor positive, HER2 negative Breast Cancer.
2. Age: 18 - 75 years old, postmenopausal women or prepostmenopausal women
3. Received prior endocrine therapy
4. One previous line of chemotherapy for advanced/metastatic disease is allowed in addition to endocrine therapy.
5. Eastern Cooperative Oncology Group [ECOG] 0-1

Exclusion Criteria:

1. Patients who received prior treatment with any CDK4/6 inhibitor, everolimus or fulvestant.
2. Clinically significant cardiovascular and cerebrovascular diseases,including but not limited to severe acute myocardial infarction within 6 months before enrollment, unstable or severe angina, Congestive heart failure (New York heart association (NYHA) class > 2), or ventricular arrhythmia which need medical intervention.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Estimated)
Dates: Start 2019-06-13 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Investigator-assessed PFS | Up to approximately 24 months.
  Investigator-assessed Progression Free Survival

SECONDARY OUTCOMES:
Progression-free Survival (PFS) per RECIST 1.1 | Up to approximately 24 months.
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on blinded independent central review or death due to any cause, whichever occurs first.
OS | Up to approximately 2 years
  Overall Survival
ORR | Up to approximately 24 months.
  Objective Response Rate
DoR | Up to approximately 24 months
  Duration of Objective Response
CBR | Up to approximately 24 months.
  Clinical Benefit rate
AEs and SAEs | Up to approximately 24 months.
  Number of Participants With adverse events (AEs) and serious adverse events (SAEs) Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v4.03.
Ctrough | Up to 4 weeks
  Ctrough

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Science, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu YP, Hu MH, Lin PP, Li T, Liu SQ, Wang YY, Li SR, Li XK, Wang CJ, Cao Y. Evaluation of the Effect of Food on the Pharmacokinetics of SHR6390, An Oral CDK4/6 Inhibitor, in Healthy Volunteers. Drugs R D. 2022 Jun;22(2):175-182. doi: 10.1007/s40268-022-00390-7. Epub 2022 May 30. PMID 35635717
- [Derived] Xu B, Zhang Q, Zhang P, Hu X, Li W, Tong Z, Sun T, Teng Y, Wu X, Ouyang Q, Yan X, Cheng J, Liu Q, Feng J, Wang X, Yin Y, Shi Y, Pan Y, Wang Y, Xie W, Yan M, Liu Y, Yan P, Wu F, Zhu X, Zou J; DAWNA-1 Study Consortium. Dalpiciclib or placebo plus fulvestrant in hormone receptor-positive and HER2-negative advanced breast cancer: a randomized, phase 3 trial. Nat Med. 2021 Nov;27(11):1904-1909. doi: 10.1038/s41591-021-01562-9. Epub 2021 Nov 4. PMID 34737452